CLINICAL TRIAL: NCT04605679
Title: Transplantation of HCV Donor Kidneys in HCV Negative or Previously Successfully Treated Recipients
Brief Title: Hepatitis C Virus (HCV) Positive Kidney Grafts in HCV Negative Recipients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5200098
Record Dates: First submitted 2020-10-25; First posted 2020-10-28 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Kidney Failure
Keywords: HCV
MeSH Terms: conditions — Renal Insufficiency | interventions — Kidney Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recipient of HCV positive kidney graft (Experimental): A single center, open-label, pilot study examining 20 adult HCV negative kidney transplant patients who receive an HCV infected graft. Target start date for antiviral therapy will be within 3 months after kidney transplantation, unless extenuating clinical circumstances arise (such as the development of fibrosing cholestatic HCV, which would prompt earlier treatment, or clinical events or comorbidities which would prompt delay in treatment).
  Interventions: Procedure: Kidney Transplantation

INTERVENTIONS:
Procedure: Kidney Transplantation — A HCV negative or previously successfully treated recipient with a HCV positive kidney graft

SUMMARY:
To determine the efficacy and safety of transplanting HCV positive kidney allografts to HCV sero-negative patients who are on the waiting list.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18 and older
* English and Spanish speaking patients
* Active on the waiting list for kidney transplantation
* Donor organ with Antibody and NAT (nucleic acid test) positive for HCV
* HCV negative recipient; this includes patients who never had HCV and those with HCV previously eradicated with antiviral therapy. The latter is defined as those with undetectable HCV viral load at least 3 months since stopping therapy.
* Willing and able to provide written informed consent

Exclusion Criteria:

* Participants co-infected with HIV
* Donor previously treated with an NS5a containing regimen (if treatment history of donor known)
* Known allergies or hypersensitivity to DAA or RBV
* Pregnancy and/or actively breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
1-year graft and patient survival | From the date of transplant through the last day of 12 month post transplant
  Will track subjects post transplant for 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael E de Vera, MD, Principal Investigator — Loma Linda University Health
Locations (1):
- Loma Linda University Health-Transplant Institute, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reese PP, Abt PL, Blumberg EA, Van Deerlin VM, Bloom RD, Potluri VS, Levine M, Porrett P, Sawinski D, Nazarian SM, Naji A, Hasz R, Suplee L, Trofe-Clark J, Sicilia A, McCauley M, Gentile C, Smith J, Niknam BA, Bleicher M, Reddy KR, Goldberg DS. Twelve-Month Outcomes After Transplant of Hepatitis C-Infected Kidneys Into Uninfected Recipients: A Single-Group Trial. Ann Intern Med. 2018 Sep 4;169(5):273-281. doi: 10.7326/M18-0749. Epub 2018 Aug 7. PMID 30083748
- [Background] Durand CM, Bowring MG, Brown DM, Chattergoon MA, Massaccesi G, Bair N, Wesson R, Reyad A, Naqvi FF, Ostrander D, Sugarman J, Segev DL, Sulkowski M, Desai NM. Direct-Acting Antiviral Prophylaxis in Kidney Transplantation From Hepatitis C Virus-Infected Donors to Noninfected Recipients: An Open-Label Nonrandomized Trial. Ann Intern Med. 2018 Apr 17;168(8):533-540. doi: 10.7326/M17-2871. Epub 2018 Mar 6. PMID 29507971
- See also: Twelve-Month Outcomes After Transplant of Hepatitis C-Infected Kidneys Into Uninfected Recipients — https://pubmed.ncbi.nlm.nih.gov/30083748
- See also: Direct-Acting Antiviral Prophylaxis in Kidney Transplantation From Hepatitis C Virus-Infected Donors to Noninfected Recipients — https://pubmed.ncbi.nlm.nih.gov/29507971